CLINICAL TRIAL: NCT04622215
Title: Diuresis, Functional Bladder Capacity and LUTS (Lower Urinary Tract Symptoms) in CKD (Chronic Kidney Disease) and ESRD (End Stage Renal Disease) Patients.
Brief Title: Diuresis, Functional Bladder Capacity and LUTS in CKD and ESRD Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018-284
Record Dates: First submitted 2018-12-05; First posted 2020-11-09 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2018-10

CONDITIONS: Lower Urinary Tract Symptoms; End Stage Renal Disease
Keywords: Lower Urinary Tract Symptoms; End Stage Renal Disease
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICIQ questionnaire (Other)
  Interventions: Diagnostic Test: ICIQ questionnaire

INTERVENTIONS:
Diagnostic Test: ICIQ questionnaire — questionnaire

SUMMARY:
The aim of the study is to evaluate the prevalence of LUTS in patients with moderate to severe (Stage IIIb), severe (Stage IV) CKD and ESRD : Stage V CKD) without renal transplantation (both pre-dialysis and dialysis patients). The study will also investigate the correlation between the diuresis, functional bladder capacity and LUTS in this population.

By means of the obtained results, the investigators hope to be able to predict at which values of diuresis and functional bladder capacity these patients will start to develop LUTS. The investigators will also evaluate the impact of LUTS on the quality of life of these patients.

DETAILED DESCRIPTION:
Pre-dialysis and peritoneal dialysis (home dialysis) and hemodialysis patients will be asked to fill in a 24h voiding diary the day prior to the control visit or dialysis session, or this can be registered the day of planned 24h urine collection.

All patients will be asked to fill a ICIQ-LUTS questionnaire. The ICIQ-LUTS questionnaire is a validated questionnaire to investigate the presence of LUTS in a non-invasive way: ICIQ-FLUTS(female lower urinary tract symptoms) for female patients and ICIQ-MLUTS(male lower urinary tract symptoms) for male patients.

Following patient data will be registered:

* Age
* Gender
* eGFR(estimated Glomerular Filtration Rate) (CKD-EPD)
* Cause of CKD-ESRD
* In case of dialysis: duration modality (hemodialysis or peritoneal dialysis)
* Antecedents
* Comorbidities
* Medication
* 24h voiding diary
* LUTS questionnaire

ELIGIBILITY:
Inclusion Criteria:

* >18years old
* GFR(CKD-Epi) < 45 ml/min and persisting minimal diuresis
* able to read and understand Dutch, French or English

Exclusion Criteria:

* <18 years old
* eGFR (CKD-EPI) > 45 ml/min
* eGFR (CKD-EPI) < 45 ml/min and > 3 months absent persisting minimal diuresis
* unable to read and understand Dutch, French or English
* renal transplant recipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
prevalence of LUTS in ESRD by ICIQ questionnaire | up to 6 month
  A ICIQ male or female LUTS questionnaire will be taken by investigator in all patient who signed IC.

SECONDARY OUTCOMES:
evaluation of bladder capacity in ESRD | up to 6 month
  Patient will be asked to keep an 24hour voiding diary This consist in keeping a record of the time of voiding and the volume of urine passed in ml each void. This will be measured in milliliter

CONTACTS AND LOCATIONS:
Overall Officials: veerle de boe, md, Principal Investigator — universitair ziekenhuis VUB
Locations (3):
- Belgium (3):
  - Valida, Brussels, Brussels Capital
  - universitair ziekenhuis VUB, Jette, Vlaams Brabant
  - AZ Jan Portaels, Vilvoorde, Vlaams Brabant